CLINICAL TRIAL: NCT00272480
Title: Zidovudine Plus Lamivudine in HTLV-I-associated Myelopathy: a Randomised Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BRIDGE1.0
Record Dates: First submitted 2006-01-04; First posted 2006-01-06 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: HTLV-I-associated Myelopathy
Keywords: HAM/TSP; HTLV-I-associated myelopathy; zidovudine; lamivudine; antiretroviral therapy
MeSH Terms: conditions — Paraparesis, Tropical Spastic | interventions — lamivudine, zidovudine drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo in HAM/TSP 24
  Interventions: Drug: Placebos
- Zidvoudine plus lamivudine (Active Comparator): Zidvoudine plus lamivudine in HAM/TSP 24
  Interventions: Drug: Zidovudine/lamivudine

INTERVENTIONS:
Drug: Zidovudine/lamivudine
  Arms: Zidvoudine plus lamivudine
Drug: Placebos
  Arms: Placebo

SUMMARY:
To determine whether the use of two antiviral agents in combination will be better than placebo in the treatment of an inflammatory sidease of the spinal cord caused by HTLV-I

DETAILED DESCRIPTION:
Randomised, double-blind, placebo-controlled two centre study of zidvoudine plus lamivudine in HAM/TSP 24 patients randomised 1:1 2-4 week lead-in 6 months randomised phase followed by 6 months open-label therapy with active drug Primary endpoint: clinical Secondary endpoints: virological and immunological

ELIGIBILITY:
Inclusion Criteria:

* HTLV-I-associated myelopathy

Exclusion Criteria:

* prior exposure to zidovudine or lamivudine on disease modifying therapy
* under age 16

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 1999-11-08 (Actual); Primary Completion 2002-07-30 (Actual); Study Completion 2002-07-30 (Actual)

PRIMARY OUTCOMES:
Timed walk | 6 months
  Time taken to walk 13m
Osame's Motor Disability Score | 6 months
  0 - 4 (Unaided walk), 5 - 8 (Needs aid to walk), 9 - 13 (Unable to walk)
Pain score | 6 months
  11 point Visual Analogue Scale 0 = no pain, 10 = worse pain
Urinary frequency | 6 months
  Number of times passing urine during the daytime
HTLV-1 proviral load | 6 months
  The number of copies of HTLV DNA in 100 peripheral blood mononuclear cells

SECONDARY OUTCOMES:
CD25% | 6 months
  Expression of CD25 on T-cells
HLA-DR% | 6 months
  Expression of HLA-DR on T-cells

CONTACTS AND LOCATIONS:
Overall Officials: Graham P Taylor, FRCP, Principal Investigator — Imperial College London
Locations (1):
- Imperial College, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taylor GP et al The Bridge Study - A double-blind, placebo controlled trial of zidovudine plus lamivudine for the treatment of patients with HTLV-I-associated myelopathy AIDS Research and Human Retroviruses 2003;19 (suppl 1) #O23
- [Result] Taylor GP, Goon P, Furukawa Y, Green H, Barfield A, Mosley A, Nose H, Babiker A, Rudge P, Usuku K, Osame M, Bangham CR, Weber JN. Zidovudine plus lamivudine in Human T-Lymphotropic Virus type-I-associated myelopathy: a randomised trial. Retrovirology. 2006 Sep 19;3:63. doi: 10.1186/1742-4690-3-63. PMID 16984654